CLINICAL TRIAL: NCT06468527
Title: A Phase IIb, Multicentre, Randomised, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Efficacy and Safety of Dirocaftor/Posenacaftor/Nesolicaftor in Subjects With Cystic Fibrosis Aged 18 Years or Older
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of Dirocaftor/Posenacaftor/Nesolicaftor in Adults With CF
Acronym: CHOICES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kors van der Ent (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor-Investigator, Kors van der Ent, Project Leader and Coordinating Investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIT-CF-001
Record Dates: First submitted 2024-06-03; First posted 2024-06-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CFTR modulator; Intestinal organoids
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diponecaftor/Placebo (Other): Diponecaftor once daily for 8 weeks followed by placebo once daily for 8 weeks. In between both periods there will be a washout period to minimize a possible carryover effect.
  Interventions: Drug: Diponecaftor; Drug: Placebo
- Placebo/Diponecaftor (Other): Placebo once daily for 8 weeks followed by diponecaftor once daily for 8 weeks. In between both periods there will be a washout period to minimize a possible carryover effect.
  Interventions: Drug: Diponecaftor; Drug: Placebo

INTERVENTIONS:
Drug: Diponecaftor — Diponecaftor is a triple combination of DIR/POS/NES. The combination therapy will be administered orally during 8 weeks. The daily dose contains:
  * DIR 300 mg/day
  * POS 600 mg/day
  * NES 10 mg/day
Drug: Placebo — Placebo once daily for 8 weeks. Oral administration.

SUMMARY:
CF is caused by mutations in the gene that encodes the 'Cystic Fibrosis Transmembrane Conductance Regulator (CFTR)' channel. To re-establish the function of this complex chloride channel, typically two to three drug modes of action are needed. To date, clinical studies of CFTR modulators have focused on patients carrying the F508del CFTR mutation, which is present in approximately 80% of CF patients, or gating mutations which are present in 5% of CF patients (gating mutations result in a reduced opening of the CFTR-channel at the cell surface which limits the flow of chloride ions through the CFTR channel). Although CF is a monogenetic disease, the 15% remaining patients represent more than 2000 different rare and mostly uncharacterized CFTR mutations. Multiple pharma companies have one or more CF drugs in their developmental pipeline. However, it is not known which patients may respond to the drugs in the pipeline. It is hypothesized that by using individual patient's intestinal organoids to screen for drug response, a subset of patients with rare CFTR mutations can be identified who will clinically respond to drugs in the developmental pipeline. The Human Individualized Therapy of CF (HIT-CF) project has been designed to further evaluate this hypothesis. The project has received funding from the European Union's Horizon 2020 research and innovation program under grant agreement No 755021. The core of the project consists of a two-step approach to identify patients outside the existing drug label who may also benefit from CFTR-modulator treatment. In the first step of the project (HIT-CF Organoid Study, NTR7520), novel CFTR modulators and their combinations were tested on organoids from over 500 European and Israeli CF patients with rare CFTR mutations to identify patients who are predicted to clinically benefit from these treatments. The second step will evaluate the predicted clinical effect of the CFTR modulators in subjects identified by their organoid response to investigational products. CFTR modulators from the HIT-CF participating pharmaceutical company, FAIR Therapeutics, will be evaluated in the CHOICES clinical study described in this protocol. Data from this clinical study will be compared with the HIT-CF Organoid Study results to validate the organoid model.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet ALL the following criteria in order to participate:

1. Male or female subjects who completed the HIT-CF Organoid Study and are 18 years of age or older on the date of informed consent
2. Confirmed diagnosis of CF as follows:

   * Sweat chloride value of ≥60 mmol/L based on quantitative pilocarpine iontophoresis (at screening) OR 2 CF-causing mutations AND
   * chronic sinopulmonary disease or gastrointestinal/nutritional abnormalities
3. Clinically stable CF disease in the opinion of the investigator with no significant changes in health status within 28 days prior to Day 1
4. Forced expiratory volume in one second (FEV1) ≥40% of predicted to ≤90% of predicted at the Screening Visit, based on the Global Lung Function Initiative (GLI) -2012 multi-ethnic all-age reference equations
5. Body mass index (BMI) ≥16 kg/m2 and ≤30 kg/m2
6. Non-smoker and non-tobacco user (including all inhalational nicotine delivery systems) for a minimum of 30 days prior to screening, and subject agrees not to smoke or use tobacco for the duration of the study
7. Subjects of childbearing potential must meet contraception requirements (Section 13.3.1)
8. Willing to remain on a stable medication regimen for CF from 28 days before Day 1 through the last study visit
9. Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, and other study procedures
10. Selected by an unblinded coordinating team based on organoid response or random selection
11. Subject will sign and date an informed consent form (ICF

Exclusion Criteria:

A subject who meets ANY of the following criteria will be excluded from participation:

1. Subject has at least one of the following CFTR-mutations: F508del, G551D, G1244E, G1349D, G178R, G551S, S1251N, S1255P, S549N, S549R, R117H, A455E, 3849+10kbC>T OR A combination of any two of the following mutations: any nonsense mutation, 1717-1G>A, 621+1G>T, 3120+1G>A, 1898+1G->A, CFTRdele2,3, and 2183AA->G
2. History or current evidence of any clinically significant cardiac (eg, heart failure, left ventricular hypertrophy, myocardial infarction, and arrhythmia), endocrinologic, hematologic, hepatobiliary (eg, clinically significant cirrhosis with or without portal hypertension, hepatitis B or hepatitis C), immunologic, metabolic, urologic, pulmonary (besides CF), neurologic (eg, subarachnoid haemorrhage, intracranial haemorrhage, cerebrovascular accident, intracranial trauma, and autonomic neuropathy), dermatologic, psychiatric, renal, or other major disease, that is unstable or could interfere with the subject's participation in or completion of the study, in the opinion of the investigator
3. Clinically significant screening results that would exclude subject from the study (eg, medical history, physical examination, ECG, vital sign, pulse oximetry, and laboratory profiles) or any conditions that, would make the subject unsuitable for enrolment or could interfere with the subject's participation in or completion of the study, in the opinion of the investigator. The medical monitor must be contacted for review of any subjects with screening results or conditions that may make them unsuitable for enrolment or could interfere with participation in or completion of the study.
4. Prolonged QTcF >450 msec at screening
5. Abnormal liver function as defined by AST, ALT, gamma-glutamyl transferase (GGT), or alkaline phosphatase ≥3 times or total bilirubin ≥2 times upper limit of the normal range
6. Haemoglobin <10 g/dL
7. Platelet count <150,000 cells/mm3
8. Abnormal renal function at screening defined as creatinine clearance <60 mL/min using the Modified Diet in Renal Disease (MDRD)
9. Hospitalisation, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness (in the opinion of the investigator) requiring an increase or addition of medication, such as antibiotics or corticosteroids, within 28 days of Day 1
10. Lung infection with organisms associated with a more rapid decline in pulmonary status (eg, Burkholderia cenocepacia, Burkholderia dolosa, and Mycobacterium abscessus). Subjects who have a current or past history of a positive culture must be reviewed with the medical monitor to confirm clinical stability.
11. Subject is currently taking or has taken a CFTR modulator within 28 days prior to Day 1
12. Participation in another clinical trial or treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to screening. The duration of the elapsed time may be longer if required by local regulations
13. History of cancer (excluding cervical carcinoma in situ and non-melanoma skin cancer with curative therapy for at least 5 years prior to screening)
14. History of organ or hematologic transplantation
15. History or current evidence of alcohol or drug abuse or dependence within 12 months of screening, in the opinion of the investigator
16. Initiation of any new chronic therapy (eg, ibuprofen, hypertonic saline, azithromycin, dornase alfa, aztreonam for inhalation solution, and tobramycin) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days prior to Day 1
17. Known or suspected hypersensitivity or idiosyncratic reaction to the study drugs or any components thereof
18. Pregnant or nursing women
19. Special or vulnerable status (e.g. institutionalized, or person related to or an employee of the sponsor, FAIR Therapeutics, or investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Mean percent predicted forced expiratory volume in 1 second (ppFEV1) | Measurements taken at 4, 6 and 8 weeks of treatment
  The primary endpoint in both groups is the mean percent predicted forced expiratory volume in 1 second (ppFEV1) of measurements taken after 4, 6 and 8 weeks of treatment. Period baseline values will be corrected for in the analysis.

SECONDARY OUTCOMES:
Sweat chloride | Measurements taken at 4, 6 and 8 weeks of treatment
  The average of the sweat chloride measurements taken after 4, 6 and 8 weeks of treatment.
Body weight | Measurements taken at 4, 6 and 8 weeks of treatment
  The average of the body weight measurements taken after 4, 6 and 8 weeks of treatment
Cystic Fibrosis Questionnaire Revised (CFQ R) respiratory domain | Measurements taken at 4, 6 and 8 weeks of treatment
  The average of the Cystic Fibrosis Questionnaire Revised (CFQ R) respiratory domain measurements taken after 4, 6 and 8 weeks of treatment. Scores range from 0 to 100, with higher scores indicating better health.
Safety and tolerability assessments | Through study completion, an average of 30 weeks
  Safety and tolerability assessments based on treatment-emergent Adverse Events (AEs)
Safety and tolerability assessments | Through study completion, an average of 30 weeks
  Safety and tolerability assessments based on treatment-emergent Serious Adverse events (SAEs)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Platelet count
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Liver function (total bilirubin)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Liver function (alkaline phosphatase (ALP))
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Liver function (alanine transaminase (ALT))
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Liver function (gamma-glutamyl transferase (GGT))
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Anemia (Haemoglobin (Hb))
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Anemia (Haematocrit)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Anemia (Red blood cell count)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  White blood cell count (including differential)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Glucose measured in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Sodium in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Cholesterol in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Total protein in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Potassium in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Chloride in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Bicarbonate in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Lactate dehydrogenase in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Albumine in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Calcium in blood
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  GFR MDRD (equation based on sex, ethnicity, age, blood urea nitrogen (BUN), creatinine)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Ketonuria (ketones measured by urine dipstick)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Proteinuria (protein measured by urine dipstick)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Hematuria (blood measured by urine dipstick)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Glucosuria (glucose measured by urine dipstick)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  pH of urine (pH measured by urine dipstick)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Specific gravitiy of urine (measured by urine dipstick)
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Coagulation (activated partial thromboplastin time (aPTT))
Safety and tolerability assessments | Measurement taken at 4, 6 and 8 weeks of treatment
  Coagulation (prothrombin time international normalized ratio (PT-INR))
Safety and tolerability assessments | Measurement taken at 4 weeks of treatment
  ECG QT Interval
Safety and tolerability assessments | Measurement taken at start of treatment and at 4, 6 and 8 weeks of treatment
  Systolic and diastolic blood pressure
Safety and tolerability assessments | Measurement taken at start of treatment and at 4, 6 and 8 weeks of treatment
  Heart rate
Safety and tolerability assessments | Measurement taken at start of treatment and at 4, 6 and 8 weeks of treatment
  Respiratory rate
Safety and tolerability assessments | Measurement taken at start of treatment and at 4, 6 and 8 weeks of treatment
  Body temperature
Safety and tolerability assessments | Measurement taken at start of treatment and at 4, 6 and 8 weeks of treatment
  Pulse oximetry measurements

CONTACTS AND LOCATIONS:
Overall Officials: C.K. van der Ent, Principal Investigator — UMC Utrecht
Locations (16):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium
- France (2):
  - CHU de Nice, Nice
  - Hôpital Larrey CHU Toulouse, Toulouse
- Germany (2):
  - Charité Universitätsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
- Italy (4):
  - Instituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambino Gesù, Rome
  - Azienda Ospedaliera Universitaria Integrata, Verona
- UMC Utrecht, Utrecht, Utrecht, Netherlands
- Hospital de Santa Maria, Lisbon, Portugal
- Hospital Vall d'Hebron, Barcelona, Spain
- Sahlgrenska University Hospital, Gothenburg CF center, Gothenburg, Sweden
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Brompton Hospital, London
  - University Hospital Southampton, Southampton